CLINICAL TRIAL: NCT05836272
Title: Early Administration of Norepinephrine in Sepsis (Tunisian Multicenter Randomized Trial)
Brief Title: Early Administration of Norepinephrine in Sepsis
Acronym: EA-NE-TUN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Ahlem Trifi, Associate Professor, Tunis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tunisian ICUs association
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Sepsis, Severe
Keywords: sepsis; septic shock; Norepinephrine; volume expansion; mortality
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Norepinephrine

STUDY DESIGN:
Intervention Model Description: This involves randomizing 2 independent groups according to a succession of six blocks of random permutations and this will be carried out using a computer-generated tool: the NE group (early noradrenaline group) which will receive NA at start for correction of hypotension and Placebo group (standard treatment group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early NE (Active Comparator): The early NE arm will receive low-dose NE as soon as hypotension secondary to sepsis is observed in addition to a classic therapeutic regimen that complies with the guidelines of the 2021 Surviving Sepsis Compaign. Sepsis is defined according to the sepsis 3 consensus by a sepsis related organ failure assessment (SrOFA) score greater than 2 following an infection (documented or suspected)
  Interventions: Drug: Norepinephrine Bitartrate
- Placebo (Placebo Comparator): The placebo arm will receive only the classic therapeutic regimen that complies with the guidelines of the 2021 Surviving Sepsis Compaign.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Norepinephrine Bitartrate — The NE will be prepared as follows: 4 mg mixed with 250 ml of 5% glucose resulting in a final norepinephrine concentration of 0.016 mg/ml. For the control group placebo: 250 ml of 5% glucose will be prepared.
  Both drugs will be infused via a peripheral line or a venous catheter. The intravenous infusion rate varies from 8 to 15 ml/hour, adjusted according to body weight to obtain norepinephrine at 0.05 microgram/kg/min (ie 0.128 to 0.24 mg per hour) in continuous infusion.
  Other Names: Norepinephrine 0,016 mg/ml
  Arms: Early NE
Other: Placebo — For the control group placebo: 250 ml of 5% glucose will be prepared and will be infused via a peripheral line or a venous catheter. The intravenous infusion rate varies from 8 to 15 ml/hour.
  Arms: Placebo

SUMMARY:
The management of septic states includes, in addition to the specific treatment (antimicrobials and eradication of the source), a restoration of the hemodynamic disorders and assistance of the failing organs. In general, the restoration of hemodynamic disorders begins first with volume expansion, followed by the use of Noepinephrine (NE) when the target mean arterial pressure (MAP) is not reached after optimizing the intravascular volume. Recently, several studies have supported the interest of early NE on MAP, cardiac output and mortality. It is therefore tempting to restrict fluid administration even in the initial phase of hemodynamic management of severe sepsis by starting NE earlier.

DETAILED DESCRIPTION:
Sepsis is characterized by systemic inflammation induced by a severe infection resulting in an inappropriate host response against that infection. On the microcirculatory scale, vasoplegia with capillary leakage is distinguished. Management of sepsis includes, in addition to specific treatment which includes antimicrobials and eradication of the source, restoration of hemodynamic disorders and assistance to failing organs. In general, the restoration of hemodynamic disorders begins first with volume expansion, followed by the use of vasopressors (mainly norepinephrine: NE as first-line therapy) when the mean arterial pressure target (MAP: reflecting the perfusion pressure organs) is not reached after optimizing the intravascular volume.

Recently, several studies have supported the benefit of administering NE at the start of resuscitation of sepsis. Indeed, its administration at an earlier phase than usually recommended improved MAP and cardiac output with a favorable effect on mortality. At a median interval of 1.3 hours from ICU admission and exclusive administration of NE, MAP was adequately restored within a relatively short time (30 min) and was associated with a better survival rate than that predicted by the severity scores of similar patients from other series reported in the literature. In the recent Thai "CENSER" trial, shock was controlled in 76% of patients in the early NE group versus 48% (p<0.001). On the other hand, the administration of a large quantity of fluids inevitably increases the risk of fluid overload, which is a frequent complication in septic patients. In front of all these arguments, it is therefore tempting to restrict fluid administration even to the initial phase of the hemodynamic management of sepsis by starting NE earlier.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* The patient or his/her legal representative has given informed consent in writing.
* Diagnosis of sepsis according to the definitions updated by the consensus of sepsis 3.
* Mean arterial pressure < 65 mmHg

Exclusion Criteria:

* Diagnosis of septic shock prior to randomization (where NA requirements exceed those of the trial protocol)
* Pregnancy,
* Need for immediate surgery,
* Neoplasia at an advanced stage
* Circumstances where water restriction is the rule:
* Acute pulmonary edema
* Acute coronary syndrome,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
shock control | within 6 hours
  shock control is defined by a composite criterion (MAP > 65 mm Hg for 2 consecutive measurements and urinary output > 0.5 ml/kg/h for 2 consecutive hours)

SECONDARY OUTCOMES:
Decrease in serum lactate | within 6 hours
  Decrease in serum lactate > 10% from baseline
Volume of fluid | within 48 hours
  Quantity of intravenous fluid received
Mortality | 28 days
  Mortality

OTHER OUTCOMES:
Use of invasive ventilation | 48 hours
  Use of invasive ventilation
Variation of cardiac output | Within 6 hours
  Variation of Cardiac output assessed xith transthoracic cardiac ultrasound (the 15% threshold is considered to define an increase in CO).

CONTACTS AND LOCATIONS:
Overall Officials: Ahlem Trifi, Principal Investigator — Hopital La Rabta
Locations (1):
- intensive care unit of the University Hospital Center La Rabta, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Permpikul C, Tongyoo S, Viarasilpa T, Trainarongsakul T, Chakorn T, Udompanturak S. Early Use of Norepinephrine in Septic Shock Resuscitation (CENSER). A Randomized Trial. Am J Respir Crit Care Med. 2019 May 1;199(9):1097-1105. doi: 10.1164/rccm.201806-1034OC. PMID 30704260
- [Derived] Trifi A, Abdellatif S, Mehdi A, Messaoud L, Seghir E, Mrad N, Ben Khelil J, Ben Ismail K, Merhaben T, Fradj H, Mokline A, Messaadi AA, Khiari H, Garbaa Y, Borsali Falfoul N, Ennouri E, Toumi R, Boussarsar M, Jaoued O, Atrous S, Ghezala HB, Brahmi N, Trabelsi I, Ghadhoune H, Bradaii S, Bahloul M, Ammar R, Kaaniche FM. Early administration of norepinephrine in sepsis: Multicenter randomized clinical trial (EA-NE-S-TUN) study protocol. PLoS One. 2024 Jul 18;19(7):e0307407. doi: 10.1371/journal.pone.0307407. eCollection 2024. PMID 39024364